CLINICAL TRIAL: NCT02269540
Title: A New Biomarker-Based Approach Towards Developing Improved Treatment for Major Depressive Disorder (MDD) Based Upon Targeting Monoamine Oxidase A (MAO-A)
Brief Title: A New Treatment Approach for Major Depressive Disorder Based Upon Targeting Monoamine Oxidase A (MAO-A)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Jeff Meyer, Canada Research Chair, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 137/2013
Record Dates: First submitted 2014-08-11; First posted 2014-10-21 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline; Citalopram; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sertraline and n-acetylcysteine (Experimental): Sertraline and n-acetylcysteine for seven weeks of treatment
  Interventions: Drug: Sertraline; Drug: N-acetylcysteine (NAC)
- Citalopram and n-acetylcysteine (Experimental): Citalopram and n-acetylcysteine for seven weeks of treatment
  Interventions: Drug: Citalopram; Drug: N-acetylcysteine (NAC)
- Existing medication treatment & NAC (Experimental): Existing depression medication treatment and n-acetylcysteine for seven weeks of treatment
  Interventions: Drug: N-acetylcysteine (NAC); Drug: Existing depression medication treatment

INTERVENTIONS:
Drug: Sertraline — selective serotonin reuptake inhibitor
  Other Names: Zoloft
  Arms: Sertraline and n-acetylcysteine
Drug: Citalopram — selective serotonin reuptake inhibitor
  Other Names: Celexa
  Arms: Citalopram and n-acetylcysteine
Drug: N-acetylcysteine (NAC) — natural health product
Drug: Existing depression medication treatment — Continuation of depression medication treatment already taken prior to study enrollment except for drugs with affinity for MAO-A or potentially influencing MAO-A levels, including phenelzine, tranylcypromine, moclobemide, cytomel and lithium
  Arms: Existing medication treatment & NAC

SUMMARY:
The investigators will be looking at MAO-A density before and after seven weeks of treatment with an antidepressant and dietary supplement. MAO-A is an enzyme that breaks down brain chemicals that regulate mood. MAO-A density is elevated in patients with major depressive episodes (MDE) secondary to major depressive disorder (MDD). Many remain treatment resistant with common antidepressant treatments and we think it may be due to poor targeting of brain pathologies. We want to test if adding a dietary supplement may normalize MAO-A.

DETAILED DESCRIPTION:
All subjects are getting the combined treatment of a selective serotonin reuptake inhibitor and the dietary supplement. There are two possible selective serotonin reuptake inhibitor treatments but the dietary supplement remains the same. No subjects are receiving the selective serotonin reuptake inhibitor alone and no subjects are receiving the dietary supplement alone. The dietary supplement is called n-acetylcysteine.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of current major depressive episode and major depressive disorder
* Hamilton Depression Rating Scale score of at least 20

Exclusion Criteria:

* Comorbid axis I or II disorders
* Antidepressant use in past 6 months
* Current use of herbal remedies
* Cigarette smoking
* Drug or medication use within past 8 weeks
* History of substance abuse/neurotoxin use
* History of psychotic symptoms
* History of CNS medical illness
* Current substance use
* Test positive on pregnancy test (women)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
MAO-A distribution volume with positron emission tomography | before and after treatment, 7 weeks on average between measures
  Treatment take 1 week for titration and 6 weeks at full dose=7weeks average

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale Score | before and after treatment, 7 weeks on average between measures
  Treatment takes 1 week for titration and 6 weeks at full dose=7 weeks average
Magnetic Resonance Spectroscopy (n-acetylaspartate and glutathione levels) | before and after treatment, 7 weeks on average between measures
  Treatment takes 1 week for titration and 6 weeks at full dose=7 weeks average
Blood markers of monoamine oxidase-A fragment level and glutathione level | before and after treatment, 7 weeks on average between measures
  Treatment takes 1 week for titration and 6 weeks at full dose=7 weeks average

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Meyer, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health; University of Toronto
Locations (1):
- Research Imaging Centre, Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research